CLINICAL TRIAL: NCT00899600
Title: Intra-operative Ketamine Infusions in Patients With Chronic Lower Back Discomfort Undergoing Laminectomies.
Brief Title: Intra-operative Ketamine Infusions in Opioid-dependent Patients With Chronic Lower Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 100674
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Results first posted 2013-04-11 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-09

CONDITIONS: Chronic Low Back Pain
Keywords: chronic pain; back surgery; opioid dependent; NMDA receptor antagonism; Ketamine; Central sensitization
MeSH Terms: conditions — Chronic Pain | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal saline (Placebo Comparator)
  Interventions: Other: Normal saline
- Ketamine (Experimental)
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Peripheral provision of 0.5mg/kg of ketamine on induction followed by a 10mcg/kg/min infusion until surgical wound closure
  Arms: Ketamine
Other: Normal saline — Normal saline at same rate as the previously described ketamine infusion (10mcg/kg/min), same amount of ketamine/placebo syringe on induction (0.5mg/kg).
  Arms: Normal saline

SUMMARY:
Noxious stimuli occurring intraoperatively and postoperatively generate central sensitization, decreasing pain thresholds and ultimately increasing analgesic requirements. The pathophysiology of central sensitization is thought to involve excitatory amino acid receptors such as N-methyl-d-aspartate (NMDA) (1, 2). Ketamine is a N-methyl-d-aspartate (NMDA) receptor antagonist that has been shown to be useful in the reduction of acute postoperative pain and analgesic consumption in a variety of surgical interventions (3).

Spine surgery provides a unique opportunity to evaluate the preemptive and preventative impact of ketamine on the primary end points of postoperative 24 and 48 hour opioid consumption in patients with chronic pain. The goal of this double blinded, prospective, randomized placebo controlled trial is to quantify the preemptive and preventative analgesic effects of ketamine infusions in this patient population. Such insight may lead to better pain control, improved satisfaction, and ultimately a reduction in side-effects related to postoperative opioid use.

DETAILED DESCRIPTION:
Noxious stimuli occurring intra-operatively and post-operatively generate central sensitization, decreasing pain thresholds and ultimately increasing analgesic requirements. The pathophysiology of central sensitization is thought to involve excitatory amino acid receptors that have been implicated in the prolongation of painful states in animal models. The N-methyl-d-aspartate (NMDA) receptor is one such excitatory amino acid receptor (1, 2).

The underlying mechanism of central sensitization is thought to involve c-fiber associated injury occurring with incision. Crile and Wall brought about the concept that attenuation of central sensitization could be accomplished via the provision of analgesic interventions (opioids, local anesthesia) prior to the noxious insult. They termed the central sensitization attenuation preemptive analgesia. The concept of preemptive analgesia was later expanded to implicate both pre and post-incisional noxious stimuli as part of this process, resulting in studies designed to provide interventions throughout the surgical intervention (peri-procedural) (3). Reduction in analgesic requirements or pain scores for more than five half-lives (1st order kinetics) following the provision of the intervening analgesic agent peri-procedurally is now known as preventative analgesia. The term preemptive analgesia is now reserved for interventions that occur only before the noxious stimuli.

Multiple studies have investigated the concepts of preemptive analgesia and preventative analgesia by providing a variety of analgesic interventions at various times throughout the surgical insult in addition to more conventional means of anesthesia provision, including opioids, Non-Steroidal Anti-Inflammatory Drugs (NSAID)s, Cyclooxygenase-II (COX-2) inhibitors, alpha-2 agonists, and ketamine (4, 5, 6). Preemptive and preventative analgesia using a variety of pharmacological agents with at least partially known mechanisms of actions has provided some insight into potential mechanisms of central sensitization.

Ketamine is a N-methyl-d-aspartate (NMDA) receptor antagonist that has been shown to be useful in the reduction of acute postoperative pain and analgesic consumption in a variety of surgical interventions with variable routes of administration. It has also been shown to be effective in the presence and absence of opioids, suggesting that it has more than one mechanism of action in preemptive and preventative analgesia, including but not limited to decreasing central excitability, decreasing acute post-operative opioid tolerance, and a possible modulation of opioid receptors (7). Ketamine is a common anesthetic agent and has been in use since the Vietnam War. Clinically, ketamine provides pain relief with minimal respiratory depression, and at higher doses (1-2mg/kg) can induce general anesthesia while maintaining blood pressure and cardiac output.

Recently, a qualitative systematic review of the role of NMDA receptor antagonists was completed. Twenty-four studies investigating the role of ketamine met the inclusion criteria of the study, 58% of which demonstrated a preemptive or preventative analgesic effect. Patients underwent a variety of surgical procedures, both ambulatory and inpatient, and there was no obvious effect of either surgical type or dose of ketamine (range 0.15 to 1mg/kg) on the success of preventative intervention. However, the authors were unable to quantify the degree of reduction in primary end-points (opioid consumption, pain scores, both) due to variability in recording of such data. In addition, most inpatient studies were limited to abdominal procedures while the outpatient studies investigated mainly knee arthroscopies, providing no insight into the degree of impact of NMDA receptor antagonism in the setting of high pre-operative opioid tolerance combined with surgical procedures known to be associated with an invariably high degree of post-operative pain. Of note, only 1/24 studies documented a significant difference in side effects related to ketamine provision in patients who had received 20mg of epidural ketamine (7).

Laminectomy procedures provide a unique opportunity to evaluate the preemptive and preventative impact of ketamine on the primary end points of acute post-operative pain scores and opioid consumption in a patient population with opioid dependence and a high degree of post-operative and intra-operative noxious stimuli. The goal of this double blinded, randomized placebo controlled trial will be to test for the presence of, and quantify, the preemptive and preventative analgesic effects of ketamine infusions in this patient population. Such insight may lead to better pain control, improved satisfaction, and ultimately a reduction in side-effects related to post-operative opioid use including but not limited to respiratory depression, constipation, and delirium.

ELIGIBILITY:
Inclusion Criteria:

* Laminectomy procedures.
* History of chronic back pain.
* Daily opioid use.
* Capable of providing informed consent.

Exclusion Criteria:

* Intolerance/allergy to ketamine.
* Intolerance/true allergy to morphine.
* Elevated intra-ocular pressure.
* Uncontrolled hypertension.
* Elevated intra-cranial pressure.
* Any history of a psychosis.
* Pregnancy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2007-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Clark, MD, Principal Investigator — DHMC
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Background] 1. Wall PD. The prevention of postoperative pain. Pain 1988; 33: 289-90. 2. Katz J. George Washington Crile, anoci-association, and preemptive analgesia. Pain 1993;53: 243-5. 3. McQual HJ. Pre-emptive analgesia. Br J Anaesth 1992;69: 1-3. 4. Moiniche S, Kehlet H, Dahl JB. A qualitative and quantitative systematic review of preemptive analgesia for postoperative pain relief: the role of timing of analgesia. Anesthesiology 2002;96: 725-41. 5. Katz J. Pre-emptive analgesia: evidence, current status and future directions. Eur J Anaesthesiol Suppl 995;10:8-13. 6. Katz J, McCartney CJ. Update on pre-emptive analgesia. Curr Opin Anesthesiol 2002; 15: 435-41. 7. McCartney et al. A qualitative systematic review of the role of N-Methyl-D-Aspartate receptor antagonists in preventative analgesia. Anesth Analg 2004; 98: 1385-1400. 8. Wu CT, Yeh CC, Yu JC, et al. Pre-incisional epidural ketamine, morphine and bupivacaine combined with epidural and general anesthesia provides pre-emptive analgesia for upper abdominal surgery. Acta Anaesthesiol Scand 2000;44: 63-8.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted over a two-year period (February 2007 to April 2009) at Dartmouth-Hitchcock Medical Center. Approval was obtained from the Committee for Protection of Human Subjects (Lebanon, NH, United States of America). Informed patient consent was obtained from all patients.
Pre-assignment Details: Three hundred and one patients were screened. Of these patients, 165 (55%) were eligible for enrollment. Sixty-one percent of eligible patients were randomized to one of the two treatment groups. No patients enrolled in the study were excluded from the primary analysis.
Groups:
- Normal Saline: Normal saline : Normal saline at same rate as the previously described ketamine infusion (10mcg/kg/min), same amount of ketamine/placebo syringe on induction (0.5mg/kg).
Period: Overall Study
Arm/Group | Normal Saline | Ketamine
Started | 50 | 52
Completed | 50 | 52
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Saline | Ketamine | Total
Number analyzed (Participants) | 50 | 52 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 40 | 82
  >=65 years | 8 | 12 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (14.4) | 51.7 (14.2) | 51.6 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 41
  Male | 28 | 33 | 61
Region of Enrollment [Number; unit: participants]
  United States | 50 | 52 | 102

OUTCOME MEASURES:

1. Primary Outcome: Morphine Consumption in the First 48 Hours After Surgery
Description: Total morphine(mg)consumed at 48 hours.
Time Frame: 48 hours
Population: See methodology
Measure: Mean (Standard Deviation); unit: mg
Groups:
- Ketamine: Ketamine 0.5 mg/kg on induction and an infusion at 10mcg/kg/min until wound closure.
Arm/Group | Normal Saline | Ketamine
Number analyzed (Participants) | 50 | 52
mg | 309 (341) | 195 (111)

2. Secondary Outcome: Hospital Duration
Time Frame: Discharge from hospital, approximately 2 days after surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Normal Saline | Ketamine
Number analyzed (Participants) | 50 | 52
minutes | 4571 (4099) | 4364 (2296)

3. Secondary Outcome: Hemodynamic Changes - Heart Rate
Description: Hemodynamic change (Heart Rate) from baseline in the intraoperative and 48-h postoperative periods
Time Frame: Baseline, Inoperative (approximately) 48 hours
Population: Analysis included only a subgroup of participants who had not used non-steroidals (NSAIDS).
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Normal Saline | Ketamine
Number analyzed (Participants) | 47 | 37
beats per minute
  Baseline Peak Heart Rate | 77.3 (13.5) | 74 (13.9)
  Interoperative Peak Heart Rate | 91.4 (13.67) | 87.6 (13.72)
  48-hours Post Operative | 98.6 (13.4) | 99.8 (20.2)

4. Secondary Outcome: Hemodynamic Changes - Blood Pressure
Description: Hemodynamic change (Blood Pressure) from baseline in the intraoperative and 48-h postoperative periods
Time Frame: Baseline, Inoperative (approximately) 48 hours
Population: Analysis included only a subgroup of participants who had not used non-steroidals (NSAIDS).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Normal Saline | Ketamine
Number analyzed (Participants) | 47 | 37
mmHg
  Baseline systolic blood pressure | 133.8 (19.5) | 132.2 (16.9)
  Baseline diatolic blood pressure | 81.3 (12.8) | 77.3 (11.3)
  Interoperative Systolic blood pressure | 139.6 (16.7) | 139.9 (18.3)
  Interoperative diastolic blood pressure | 80.8 (13.2) | 77.8 (13.7)
  48-hours post operative systolic blood pressure | 133 (16.4) | 129.7 (12.2)
  48-hours post operative diastolic blood pressure | 75.9 (8.9) | 75.6 (8.6)

5. Secondary Outcome: Percentage of Participants With Complications/Adverse Events
Description: Adverse events
Time Frame: 48 hours and 6 weeks
Measure: Number; unit: Percent
Arm/Group | Normal Saline | Ketamine
Number analyzed (Participants) | 50 | 52
Percent
  Nausea, 48 hours | 22.5 | 26.9
  Vomiting, 48 hours | 12.2 | 15.4
  Hallucinations, 48 hours | 2.0 | 1.9
  Urinary Retention, 48 hours | 2.0 | 7.7
  Nausea, 6 weeks | 17.0 | 11.8
  Vomiting, 6 weeks | 8.5 | 9.8
  Hallucinations, 6 weeks | 23.4 | 11.8
  Urinary Retention, 6 weeks | 57.5 | 45.1

ADVERSE EVENTS:
Arm/Group | Normal Saline | Ketamine
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/52
Other Adverse Events (participants affected / at risk) | 4/50 | 5/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Saline (N=50) | Ketamine (N=52)
Nausea/vomiting during the hospital admission as reported at the 6-wk f/u visit. (Gastrointestinal disorders) | 4 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes